CLINICAL TRIAL: NCT06033118
Title: Gemox Combined With Anlotinib and Sintilimab in Advanced Combined Hepatocellular-cholangiocarcinoma: an Exploratory Study
Brief Title: Gemox Combined With Anlotinib and Sintilimab in Advanced cHCC-ICC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Director, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cHCC-ICC
Record Dates: First submitted 2023-07-10; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Combined Hepatocellular Cholangiocarcinoma
MeSH Terms: interventions — gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemox combined with Anlotinib and Sintilimab (Experimental): Gemox chemotherapy（gemcitabine 1g/m2 ivgtt d1,d8 +oxaliplatin 85g/m2 ivgtt d1，q3w，anlotinib (8mg po d1-14 q3w )and Sintilimab (200mg ivgtt d1 q3w)
  Interventions: Drug: gemcitabine ,oxaliplatin,anlotinib,Sintilimab

INTERVENTIONS:
Drug: gemcitabine ,oxaliplatin,anlotinib,Sintilimab — Gemox chemotherapy（gemcitabine 1g/m2 ivgtt d1,d8 +oxaliplatin 85g/m2 ivgtt d1，q3w，anlotinib (8mg po d1-14 q3w )and Sintilimab (200mg ivgtt d1 q3w)

SUMMARY:
The Purpose of This Study is to Evaluate the Efficacy and Safety of Gemox combined with Anlotinib and Sintilimab as first-lineTherapy for Patients With advanced combined hepatocellular-cholangiocarcinoma.

DETAILED DESCRIPTION:
Combined hepatocellular-cholangiocarcinoma (cHCC-CCA) accounts for 0.4%-14.2% of primary hepatocellular carcinoma. As imaging and pathological diagnostic techniques for liver tumors have improved, the detection rate of cHCC-CCA puncture biopsies and surgical procedures has increased. Oxaliplatin-containing chemotherapy was previously recommended for the treatment of advanced cHCC-ICC, but its efficacy was not satisfactory. Targeted therapy and immunotherapy have made breakthroughs in both advanced HCC and CCA, providing a new direction for exploration in the treatment of advanced cHCC-CCA. Currently, targeted combination immunotherapy has become the preferred first-line treatment strategy for advanced HCC. Chemotherapy combined with immunotherapy is also the preferred first-line treatment option for advanced CCA. To balance the treatment of HCC and ICC, this study further investigates the efficacy and safety of Gemox chemotherapy combined with anlotinib and Sintilimab(anti-PD-1 monoclonal antibody) immunotherapy in advanced cHCC-ICC, to provide a new treatment strategy and reference for the clinical treatment of advanced cHCC-CCA patients.

ELIGIBILITY:
Inclusion Criteria:

1. .Age 18-75 years;
2. .Histologically or cytologically confirmed diagnosis of aCombined hepatocellular-cholangiocarcinoma;
3. .Non resectable or metastatic cHCC-ICC patients who have not received systemic treatment or first-line treatment progress (only non arotinib Targeted therapy or non GEMOX chemotherapy) in the past, and have at least one measurable lesion (RECIST v1.1);
4. .Life expectancy ≥ 3 months;
5. .ECOG PS 0-1;
6. .Child Pugh A/B ≤ 7;
7. .Adequate organ function including the following:Total bilirubin ≤1.5 times upper limit of normal (ULN),Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3×ULN,Alkaline phosphatase≤2.5×ULN (If the tumor invaded the liver, ≤3×ULN), Serum creatinine≤1.5×ULN,Serum amylase and lipase≤1.5×ULN,International standardized ratio (INR)/partial prothrombin time (PTT)≤1.5×ULN;Platelet count ≥ 75,000 /mm3.Hemoglobin (Hb) ≥ 9 g/dL.Absolute neutrophil count (ANC) ≥ 1500/mm3.
8. .Strict contraception.
9. .Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Has a history of severe allergic reactions to chimeric, human or humanized antibodies, or fusion proteins.
2. Pregnant or lactating women, men and women of childbearing age who are unwilling or unable to take effective contraceptive measures;
3. History of other malignant tumors in the past 5 years, except for malignant tumors that have received treatment for the purpose of cure, and have no known active diseases for ≥ 5 years before the first administration, and have a low potential risk of recurrence; Fully treated non Melanoma skin cancer or malignant lentigo without disease evidence; Fully treated Carcinoma in situ, no disease evidence;
4. Moderate or higher amounts of pleural and ascitic fluid with clinical symptoms;
5. Active bleeding or abnormal coagulation function (PT>16s, APTT>43s, INR>1.5) × ULN), with a tendency to bleed or undergoing thrombolysis, anticoagulation, or antiplatelet therapy;
6. Hepatic encephalopathy;
7. Within the past 6 months, there has been a history of gastrointestinal bleeding or a clear tendency for gastrointestinal bleeding, such as known local active ulcer lesions, fecal occult blood+or above, which cannot be included in the group; If there is continuous fecal occult blood, gastroscopy should be performed;
8. Patients with severe gastroesophageal varices who require interventional treatment;
9. Untreated active hepatitis B. (Note: Hepatitis B patients who receive antiviral treatment and whose HBV Viral load is less than 2000IU/ml can be allowed to participate in the study)
10. Active hepatitis C, that is, those who are anti-HCV positive or HCV-RNA positive and have abnormal liver function;
11. Having a history of psychotropic substance abuse, unable to quit, or having a history of mental disorders;
12. Patients who received solid organ transplantation or bone marrow transplantation, or had active autoimmune diseases requiring systemic Sex therapy within 2 years before the first administration;
13. Existence of immune deficiency diseases or HIV infection;
14. There has been objective evidence that Pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia and serious impairment of lung function exist in the past or at present;
15. Major surgery on the liver or other parts has been performed within 4 weeks before the first administration, or minor surgery (such as simple resection, tooth extraction, etc.) has been performed within 1 week before the first administration;
16. Received the vaccine within 30 days before the first administration;
17. Abdominal fistula, gastrointestinal perforation, or abdominal abscess occurred within 4 weeks prior to the first administration;
18. For any significant clinical and laboratory abnormalities, the researchers believe that they will affect the safety evaluators, such as: active infection requiring systemic Sex therapy, uncontrollable diabetes, hypertension patients who cannot fall to the normal range (systolic pressure>140mmHg, diastolic pressure>90mmHg), myocardial infarction within 6 months, thyroid dysfunction (>NCI CTCAE v4.0 Level 1 standard) after treatment with two or less antihypertensive drugs;
19. Researchers believe that it is not suitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Every 2 cycles (each cycle is 21 days)starting from the first cycle, and every 3 cycles after 6 cycles
  Objective Response Rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1

SECONDARY OUTCOMES:
Safety and tolerability | 3 months after the last administration of drugs
  Incidence of Treatment-Emergent Adverse Events,Version 5.0 and AEs leading to dose interruption or discontinuation.
PFS | Every 2 cycles(each cycle is 21 days) starting from the first cycle, and every 3 cycles after 6 cycles
  Progression-free survival is determined from the date of treatment to PD or death from any cause
OS | Every 2 cycles(each cycle is 21 days) starting from the first cycle, and every 3 cycles after 6 cycles
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up